CLINICAL TRIAL: NCT01287078
Title: Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans Syndrome
Brief Title: Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for the Treatment of Bronchiolitis Obliterans Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110068; 11-H-0068
Record Dates: First submitted 2011-01-29; First posted 2011-02-01 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2018-08-31

CONDITIONS: Constrictive Bronchiolitis; Bronchiolitis Obliterans; Graft vs Host Disease; Bronchiolitis, Exudative; Bronchiolitis, Proliferative
Keywords: Peripheral Blood Stem Cell Transplant; Inhaled Cyclosporine; Graft-Versus-Host Disease; GVHD; Bronchiolitis Obliterans; Lung
MeSH Terms: conditions — Bronchiolitis Obliterans; Graft vs Host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inhaled Cyclosporine in Lung Transplant and HSCT Recipients (Experimental): Subjects with Bronchiolitis Obliterans Syndrome (BOS) received cyclosporine inhalation solution (CIS) 150 mg, three times weekly during weeks 1-5. Dose escalated to 300 mg three times weekly from weeks 6-8. Study drug administration ended at week 19.
  Interventions: Drug: Cyclosporine Inhalation Solution

INTERVENTIONS:
Drug: Cyclosporine Inhalation Solution — sterile, clear, colorless, preservative-free solution of cyclosporine (USP) in propylene glycol developed specifically for administration by oral inhalation.

SUMMARY:
Background:

- Bronchiolitis obliterans or bronchiolitis obliterans syndrome is a lung disorder that occurs as a complication of either lung transplantation or bone marrow/blood stem cell transplantation. One of the complications of transplant is the occurrence of graft versus host disease (in hematopoietic stem cell transplants) and host versus graft disease (in lung transplantation). In these diseases, the cells attack the lungs and cause irreversible small airway fibrosis referred to as bronchiolitis obliterans syndrome. When a patient develops fibrosis of the lungs or bronchioles, the lungs no longer work properly, which causes difficulties with breathing that lead to a diminished quality of life and an increased risk of death. Treatment typically involves immunosuppressive therapy such as oral cyclosporine or steroid therapy, but these treatments are only marginally effective and can cause significant toxicities and increase the risk of infections. Inhaled cyclosporine (CIS) achieves higher concentrations of cyclosporine in the lungs and lower concentrations of cyclosporine in the blood than oral cyclosporine. Therefore, it could have advantages over conventional oral immunosuppressive therapies used to treat this disorder. Researchers are interested in testing whether inhaled cyclosporine therapy could be used as a safe and effective treatment for bronchiolitis obliterans or bronchiolitis obliterans syndrome occurring after bone marrow/blood stem cell or lung transplants.

Objectives:

- To evaluate whether inhaled cyclosporine (CIS) can improve or stabilize lung function and quality of life in individuals with bronchiolitis obliterans.

Eligibility:

- Individuals between 10 and 80 years of age who have been diagnosed with bronchiolitis obliterans or bronchiolitis obliterans syndrome after blood or lung transplants.

Design:

* Participants will be screened with a full medical history and physical examination, as well as blood and urine tests, lung function tests, imaging studies, bronchoalveolar lavage samples, and quality of life questionnaires.
* Participants will take cyclosporine inhalation solution through a nebulizer. The nebulizer generates a mist of cyclosporine inhalation solution (CIS), which is then breathed in through a mouthpiece. The process takes approximately 20 minutes. The solution will be provided in single-use vials.
* Participants will continue to take all medications for post-transplant care as required by their doctor and the study researchers. Attempts will be made to reduce the doses and types of immunosuppressants given to participants on the study, as long as the treatment continues to produce improved or stable lung function.
* Participants will have study visits every 3 weeks with blood and urine tests, lung function tests, and imaging studies. Participants will undergo repeat bronchoalveolar sample at week 9 and 18. Participants will also complete quality of life questionnaires as directed. Treatment will continue for a minimum of 18 weeks, followed by a final follow-up visit 2 weeks after the end of the study.
* Participants who benefit from the inhaled cyclosporine (CIS) may continue to receive further therapy with inhaled cyclosporine at the end of the study by participation in a separate study extension.

DETAILED DESCRIPTION:
Bronchiolitis Obliterans (BO) is an obstructive lung disease that can affect individuals that have undergone a lung or hematopoietic stem cell transplant. BO has been studied most extensively in lung transplant recipients, where it is considered to represent chronic lung rejection. It is the leading cause of death after lung transplant, with mortality rates up to 55%. In hematopoietic stem cell transplantation, BO is thought to be a manifestation of chronic graft-vs-host disease (GVHD). Up to 45% of patients undergoing hematopoietic stem cell transplantation at the NHLBI develop a decline in pulmonary function. Conventional therapy for patients who develop BO consists of augmentation of systemic immunosuppressants. Systemic immunosuppression has limited efficacy for BO and is associated with deleterious consequences including increased risk of infections and decreased graft-versus tumor/leukemia effects.

Recently, cyclosporine inhalation solution (CIS) in solution with propylene glycol has been shown to improve overall survival and chronic rejection-free survival in lung transplant patients. These findings suggest targeted delivery of immunosuppressive therapy to the diseased organ warrants further investigation as this may minimize the morbidity associated with systemic immunosuppression. However, there currently exists limited data regarding the overall efficacy of inhaled cyclosporine to treat established BO following lung transplantation. Furthermore, inhaled cyclosporine has not been studied in the treatment of BO following hematopoietic stem cell transplantation.

Here, we propose to evaluate the safety, efficacy, and pharmacodynamics of inhaled cyclosporine for the treatment of BO. Two distinct patient populations will be offered enrollment in this protocol: hematopoietic transplant recipients with BO (group A) and lung transplant recipients with BO (group B). Study participants will receive CIS at an initial dose of 150mg, three times weekly. Patients will undergo dose titration to a maximum dose of 300mg, three times weekly. Drug deposition and pharmacokinetic analyses will be performed at the initiation of treatment. Clinical parameters, including pulmonary function tests, will be measured in addition to laboratory markers of the anti-inflammatory response to CIS. Adverse events associated with treatment will be recorded.

The primary objective is to 1) assess the safety and efficacy of inhaled cyclosporine as a new therapy in hematopoietic transplant patients and lung transplant patients with established BO. Additionally, we seek to promote a better understanding of the pathogenesis of BO in these two transplant groups and to assess the anti-inflammatory effects of inhaled cyclosporine in patients that develop this complication.

The primary endpoint of each study group is the best response, FEV1 improvement or stabilization from study baseline at week 18 for two successive measures, at least 1 week apart, no more than 2 weeks apart. Secondary endpoints include the toxicity profile as measured by CTCAE criteria (safety), the study of pharmacokinetics and lung deposition characteristics of inhaled cyclosporine, improvement in high resolution chest CT images, results of peripheral blood and bronchoalveolar cytokine arrays to assess secondary markers of inflammation, and functional capacity measurements using a six-minute walk test.

ELIGIBILITY:
* INCLUSION CRITERIA:

History of:<TAB>

-Hematopoietic stem cell transplant recipients at least 99 days post transplant (group A)

Or

* Lung transplant recipients at least 6 months post transplant (Group B)
* Biopsy proven bronchiolitis obliterans (confirmed by NIH pathology department) or Bronchiolitis Obliterans Syndrome (BOS) as defined by:
* FEV1 less than 75 percent predicted and
* No evidence of pulmonary infection as a causative etiology to lung dysfunction or other causative etiology
* Decline in FEV1 (The FEV1 values used to determine BOS will be the average of 2 measurements of FEV1 taken sequentially at least 3 weeks apart up to 6 months apart) compared to pre-transplant baseline for group A or compared to best post-transplant measurement in group B.
* For hematopoietic transplant patients, FEV1 must have declined less than 10 percent from pre-transplant baseline (group A)
* For lung transplant patients, FEV1 must have declined greater than 20 percent from best post-transplant measurement (group B)

And one of the following:

* FEV1/FVC less than 0.7
* Air trapping seen on CT scan or RV greater than 20 percent predicted
* Evidence of cGVHD affecting at least one other organ system (group A)
* Age 10-80 years
* Progressive disease or stable disease (active BOS, stable by FEV1 criteria) on immunosuppressants at study entry
* Progressive disease at study entry: Diagnosis of BO or BOS with evidence of a progressive decline in FEV1. A documented decline (greater than or equal 10 percent) in FEV1 has occurred within 18 weeks (minimum documentation of 3 weeks) preceding study enrollment
* Stable disease at study entry: Diagnosis of BO or BOS on immunosuppressive therapy with evidence of stable disease (active BOS, stable by FEV1 criteria), as documented by a stable FEV1 (increase <5% and decrease <10%) within 18 weeks (minimum documentation of 3 weeks) preceding study enrollment
* Patients on calcineurin inhibitors at study entry will be required to be on a stable dose of the calcineurin inhibitor for 4 weeks prior to study enrollment

EXCLUSION CRITERIA:

* Evidence of uncontrolled, pulmonary infection
* Patients with unstable coronary insufficiency, severe cardiac arrhythmias, and/or uncontrolled hypertension.
* History of hypersensitivity to propylene glycol
* History of allergic reaction or hypersensitivity to Technetium- 99m sulfur colloid, used in lung deposition studies
* ECOG performance status greater than or equal to 3
* Serum creatinine >2.5 mg/dl
* Documented allergy or intolerance to cyclosporine
* Patient pregnant or breast feeding or not willing to use an approved method of birth control
* Inability to comprehend the investigational nature of the study and provide informed consent
* Life expectancy less than 18 weeks.
* An increase greater than or equal to 5% and an absolute increase greater than or equal to 0.05 in FEV1 in the 18 weeks (minimum documentation of 3 weeks) preceding study enrollment
* Subjects who have had prior administration of inhaled cyclosporine.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01-29; Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole J Gormley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Afessa B, Litzow MR, Tefferi A. Bronchiolitis obliterans and other late onset non-infectious pulmonary complications in hematopoietic stem cell transplantation. Bone Marrow Transplant. 2001 Sep;28(5):425-34. doi: 10.1038/sj.bmt.1703142. PMID 11593314
- [Background] Boucek MM, Waltz DA, Edwards LB, Taylor DO, Keck BM, Trulock EP, Hertz MI; International Society for Heart and Lung Transplantation. Registry of the International Society for Heart and Lung Transplantation: ninth official pediatric heart transplantation report--2006. J Heart Lung Transplant. 2006 Aug;25(8):893-903. doi: 10.1016/j.healun.2006.05.014. No abstract available. PMID 16890109
- [Background] Savani BN, Montero A, Srinivasan R, Singh A, Shenoy A, Mielke S, Rezvani K, Karimpour S, Childs R, Barrett AJ. Chronic GVHD and pretransplantation abnormalities in pulmonary function are the main determinants predicting worsening pulmonary function in long-term survivors after stem cell transplantation. Biol Blood Marrow Transplant. 2006 Dec;12(12):1261-9. doi: 10.1016/j.bbmt.2006.07.016. PMID 17162207
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0068.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects withdrew consent after signing
Groups:
- Inhaled Cyclosporine in HSCT Recipients: Subjects who underwent Hematopoietic Stem Cell Transplant (HSCT) and developed Bronchiolitis Obliterans Syndrome (BOS) received cyclosporine inhalation solution (CIS) 150 mg, three times weekly during weeks 1-5. Dose escalated to 300 mg three times weekly from weeks 6-8. Study drug administration ended at week 19.
- Inhaled Cyclosporine in Lung Transplant Recipients: Subjects who underwent Lung Transplant (LT) and developed Bronchiolitis Obliterans Syndrome (BOS) received cyclosporine inhalation solution (CIS) 150 mg, three times weekly during weeks 1-5. Dose escalated to 300 mg three times weekly from weeks 6-8. Study drug administration ended at week 19.
Period: Overall Study
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Started | 20 | 3
Completed | 10 | 1
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients | Total
Number analyzed (Participants) | 20 | 3 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 17 | 2 | 19
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 12 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 3 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 16 | 2 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response to Treatment Based on Positive Response to Cyclosporine Inhalation Solution (CIS)
Description: Participants who responded to treatment with cyclosporine inhalation solution (CIS)
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 9 | 0

2. Primary Outcome: Overall Non-response to Treatment
Description: Participants who did not respond to treatment with cyclosporine inhalation solution (CIS)
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 7 | 2

3. Primary Outcome: Stable or Progressive Disease at Baseline With Improvement of FEV1
Description: Participants with stable or progressive disease at baseline with improvement of FEV1
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 4 | 0

4. Primary Outcome: Disease Progression at Baseline With Stablization of FEV1
Description: Participants with progressive disease at baseline with stablization of FEV1
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 2 | 0

5. Primary Outcome: Disease Stability at Baseline With Stablization in FEV1 and Greater Than 25% Decline in Systemic Immunosuppression
Description: Participants with stable disease at baseline with stablization in FEV1 and greater than 25% decline in systemic immunosuppression
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 3 | 0

6. Primary Outcome: Stable or Progressive Disease at Baseline With Greater Than 20% of Decline in FEV1
Description: Participants with stable or progressive disease at baseline with greater than 20% of decline in FEV1
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 1 | 0

7. Primary Outcome: Stable Disease at Baseline With Stablization of FEV1 and no Change or Increase in Systemic Immunosuppresion
Description: Participants with stable disease at baseline with stablization of FEV1 and no change or increase in systemic immunosuppresion
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 4 | 2

8. Primary Outcome: Disease Progression at Baseline With Decline in FEV1 Greater Than 10%
Description: Participants with progressive disease at baseline with decline in FEV1 greater than 10%
Time Frame: 18 weeks
Population: Subjects who received cyclosporine inhalation solution (CIS) for at least two weeks or three doses
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
Number analyzed (Participants) | 16 | 2
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Inhaled Cyclosporine in HSCT Recipients | Inhaled Cyclosporine in Lung Transplant Recipients
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/3
Serious Adverse Events (participants affected / at risk) | 5/20 | 0/3
Other Adverse Events (participants affected / at risk) | 18/20 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Cyclosporine in HSCT Recipients (N=20) | Inhaled Cyclosporine in Lung Transplant Recipients (N=3)
Acute myeloid leukaemia recurrent (Blood and lymphatic system disorders) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Viral pericarditis (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Cyclosporine in HSCT Recipients (N=20) | Inhaled Cyclosporine in Lung Transplant Recipients (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Dizziness (Cardiac disorders) | 1 | 0
Dyspnoea (Cardiac disorders) | 2 | 0
Oedema peripheral (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Hypoglycaemia (Endocrine disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 5 | 0
Oedema (General disorders) | 1 | 0
Graft versus host disease in eye (Immune system disorders) | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 4 | 3
Mycobacterium abscessus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 3 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Forced expiratory volume decreased (Investigations) | 0 | 1
Hyperkalaemia (Investigations) | 1 | 0
Hypernatraemia (Investigations) | 0 | 1
Hypoalbuminaemia (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neck pain (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Gait disturbance (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 1
Restlessness (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Genitourinary symptom (Renal and urinary disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oxygen saturation decreased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dizziness (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 2
Oedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT01287078/Prot_SAP_000.pdf